CLINICAL TRIAL: NCT00788099
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Plitidepsin in Combination With Sorafenib or Gemcitabine in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: Study of Plitidepsin in Combination With Sorafenib or Gemcitabine in Patients With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Pharmamar USA, Pharmamar USA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL-A-010-08
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Advanced Solid Tumors; Lymphomas
Keywords: Aplidin; Plitidepsin; Tumors; Lymphomas
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — plitidepsin; Sorafenib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Plitidepsin and Sorafenib
  Interventions: Drug: Plitidepsin and Sorafenib
- 2 (Experimental): Gemcitabine and Plitidepsin
  Interventions: Drug: Gemcitabine and Plitidepsin

INTERVENTIONS:
Drug: Plitidepsin and Sorafenib — Patients will receive i.v. plitidepsin over 1h on days 1, 8 and 15 every 4 weeks (d1, 8, 15 q4wk) and continuous oral sorafenib twice daily (bid) (a cycle is defined as an interval of 4 weeks).
  Arms: 1
Drug: Gemcitabine and Plitidepsin — Patients will receive i.v. gemcitabine over 30 minutes followed 1 hour later by plitidepsin over 1 hour on d1, 8, 15 q4wk (a cycle is defined as an interval of 4 weeks).
  Arms: 2

SUMMARY:
Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Plitidepsin in Combination with Sorafenib or Gemcitabine in Patients with Advanced Solid Tumors or Lymphomas to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of plitidepsin in combination with sorafenib or gemcitabine in patients with advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Plitidepsin in Combination with Sorafenib or Gemcitabine in Patients with Advanced Solid Tumors or Lymphomas to determine the maximum tolerated dose (MTD) and the recommended dose (RD), the pharmacokinetics (PK) of these combinations, drug-drug PK interactions, preliminary information on the clinical antitumor activity of these combinations in solid tumors,perform a preliminary pharmacogenomic (PGx) study of potential biomarkers of sensitivity/resistance to these drugs combinations and of prognostic markers of the treatment outcome in tumor tissue sample.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status (PS) of ≤ 1
* Life expectancy ≥ 3 months
* Patients with histologically/cytologically confirmed diagnosis of advanced solid tumors or lymphomas (excluding B-cell derived lineage and/or primary cutaneous and/or leukemic disease) refractory to standard therapy and with reasonable chance to benefit from any of these combinations according to the investigator's opinion.
* Patients entered at the expansion cohort of the RD must have: a) measurable disease according to RECIST, or to International Working Group Criteria (IWC) for lymphoma patients or b) Evaluable disease by serum markers in the case of prostate and ovarian cancer (according to Prostate-Specific Antigen Working Group Recommendations (PSAWGR) and Gynecologic Cancer Intergroup (GCIG) specific criteria, respectively
* At least 4 weeks since last chemotherapy (6 weeks since nitrosoureas and mitomycin C), immunotherapy or any other pharmacological treatment and radiotherapy. In the case of hormone-sensitive cancer progressing while on hormone therapy (i.e., breast, prostate cancer), hormone therapy must be either stopped 4 weeks before or continued during the trial
* Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤ 7 days before inclusion in the study): a) Platelet count ≥100 x109/L (≥ 75 x 109/L for lymphoma patients), hemoglobin ≥9.0 g/dL (≥ 8.0 g/dL for lymphoma patients) and absolute neutrophil count (ANC) ≥1.5 x109/L (≥1.0 x109/L for lymphoma patients). b) Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT): ≤ 3.0 x the upper limit of normal (ULN), independently of the presence of liver metastases. c) AP ≤2.5 x ULN (≤5 x ULN in case of extensive bone metastases). d) Total bilirubin ≤1.5 x ULN (unless due to indirect hyperbilirubinemia for the gemcitabine combination arm only). e) Calculated CrCl: ≥ 40 mL/minute (by means of Crockroft and Gault´s formula). f) CPK ≤ 2.5 x ULN. g) Albumin ≥2.5 g/dL. h) Troponin I ≤ULN
* Recovery to grade ≤1 from any AE derived from previous treatment (excluding alopecia of any grade and peripheral neuropathy ≤ grade 2)
* LVEF by ECHO or MUGA above the lower normal limit.
* Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception include complete abstinence, intrauterine device (IUD), oral contraceptive, subdermal implant and double barrier
* Voluntarily signed and dated written informed consent prior to any specific study procedure.

Exclusion Criteria:

* Previous treatment with any of the study drugs (in the expansion cohort at the RD).
* Concomitant diseases/conditions:

  * History or presence of unstable angina, myocardial infarction, valvular heart disease or congestive heart failure.
  * Previous mediastinal radiotherapy.
  * Previous treatment with doxorubicin at cumulative doses in excess of 450 mg/m2
  * Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment, and/or prolonged QT-QTc > to grade 1.
  * Active uncontrolled infection.
  * Myopathy or any clinical situation that causes significant and persistent elevation of CPK (>2.5 x ULN in two different determinations performed with one week apart).
  * Limitation of the patient's ability to comply with the treatment or follow-up protocol.
  * Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
  * Peripheral neuropathy >grade 2
* Symptomatic, progressive or requiring-corticosteroids documented brain metastases or leptomeningeal disease. Controlled and stable brain metastases without steroids are allowed
* Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding
* Patients who have had radiation therapy in greater than 35% of the bone marrow
* History of previous bone marrow and/or stem cell transplantation. (Not for patients treated at RD in the expansion cohort)
* High transfusional requirements (> 2 packages of red blood cells and/or 1 platelets transfusion) in the 30 days prior to inclusion in the study
* Participation in another clinical trial or concomitant treatment with any investigational product in the 30-day period prior to inclusion in the study.
* For sorafenib treatment only: a) Hypersensitivity to sorafenib or any component of the formulation. b) Need of chronic exposure to antacids, H-2 antagonists or proton-pump inhibitors. c) Current need for anticoagulation treatment (including low dose warfarin and LMWH treatment at full anticoagulant doses).
* Abnormal thyroid function [as per normal serum thyroid stimulating hormone (TSH) within 14 days of first dose of study treatment).
* Uncontrolled arterial hypertension (≥160/100) despite optimal medical therapy.
* Child-Pugh grade C hepatic cirrhosis of any cause
* For gemcitabine treatment only:

  * Hypersensitivity to gemcitabine or any component of the formulation.
  * Impending need for palliative radiotherapy to ameliorate painful metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of plitidepsin in combination with sorafenib or gemcitabine in patients with advanced solid tumors or lymphomas. | Along the study

SECONDARY OUTCOMES:
To characterize safety profile and feasibility, pharmacokinetics, drug-drug interactions. To obtain information on antitumor activity. | Along the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Stein, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey; Jean Charles Soria, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- The Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey, United States
- Institut Gustave Roussy, Villejuif, France